CLINICAL TRIAL: NCT03577769
Title: Health Care-associated Bacteriuria in Geriatric Wards in Strasbourg's University Hospital : a Comparative Study of Bacterial Ecology Between 2003, 2007 and 2017
Brief Title: Nosocomial Bacteriuria in Geriatric Internal Medicine Services and Follow-up Care and Geriatric Rehabilitation of the Strasbourg University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7024
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Urinary Tract Infection
Keywords: Health care associated urinary tract infection; Bacteriuria; Elderly; Geriatrics; Antimicrobial resistance; Multi-resistant bacteria
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This thesis is a comparative study of the epidemiological characteristics of health-care associated bacteriuria in short and medium term of geriatrics wards in Strasbourg's University Hospital, between 2003 and 2017, in the follow-up of Eric de Pasquale's thesis in 2010.

This comparative study will allow to see the evolution of urinary bacterial ecology, bacterial sensitivity to antibiotics, and the part of multi-resistant bacteria, during these 14 years in geriatric services in Strasbourg.

ELIGIBILITY:
Inclusion Criteria:

* patient of age who has been hospitalized in geriatric wards (rehabilitation car service and internal medicine) of Strasbourg's University hospital
* date of hospital leaving after 1/1/17 and before 1/1/18
* patient who has a health-care urinary tract infection (occurred more than 48h after admission)
* single bacteria in the CBEU
* bacteriuria > 105 cfu/mL regardless which clinical context or bacteria
* if a patient has several bacteriuria, they can be included if they appear after a precedent episode well treated or if the bacteria is different from the precedent

Exclusion Criteria:

* participation refusal
* Leaving of hospital out of the inclusion period
* Urinary tract infection which occurred less than 48h after admission (communitarian infection)
* bacteriuria < 105 cfu/mL
* multiple bacteria in the CBEU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patient of age who has been hospitalized in geriatric wards (rehabilitation car service and internal medicine) of Strasbourg's University hospital
  * date of hospital leaving after 1/1/17 and before 1/1/18
  * patient who has a health-care urinary tract infection (occurred more than 48h after admission)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial sensitivity (antibiotic resistance testing) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service Geriatrie - Soins de Suite Et Readaptation, Strasbourg, France